CLINICAL TRIAL: NCT07111494
Title: Impact of Glucagon-like Peptide-1 (GLP-1) Analogs on Disease Outcomes in Psoriatic Arthritis: A Pragmatic Randomized Controlled Trial
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Shikha Singla, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO55130
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Psoriatic Arthritis (PsA)
Keywords: Psoriatic Arthritis; GLP-1; Minimal Disease Activity; Nutrition Counseling
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Glucagon-Like Peptide-1 Receptor Agonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- GLP-1 (Active Comparator)
  Interventions: Drug: GLP-1 agonists
- Nutrition Counseling (Active Comparator)
  Interventions: Other: Nutrition Counseling

INTERVENTIONS:
Drug: GLP-1 agonists — GLP-1, any assigned drug
  Arms: GLP-1
Other: Nutrition Counseling — Nutrition Counseling in PsA
  Arms: Nutrition Counseling

SUMMARY:
Psoriatic arthritis (PsA) is a chronic inflammatory condition that affects the joints but can also have an effect on multiple parts of the body. This study will assess if the effectiveness of Glucagon-like peptide-1 (GLP-1) medications used to treat type 2-diabetes and weight management, or nutrition counseling can better treat individuals with Psoriatic Arthritis who are also needing treatment for obesity and type 2 diabetes.

The main objectives it aims to answer are:

To assess disease outcomes of PsA patients undergoing treatment for concomitant obesity and type 2 diabetes with GLP-1 analogs vs nutrition counseling.

To assess effectiveness as measured by clinical and patient reported outcome measures in patients treated with GLP-1 and nutrition counseling.

Participants will be randomized to receive a GLP-1 or nutrition counseling. Participants will be asked to come to the study center at most four times during a 24-week period. During this time participants will be asked to fill out questionnaires, receive a physical exam, and have their blood drawn.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 and older) who present to rheumatology clinic
* Participants must be able to read, understand, and provide documented informed consent as approved by the Institutional Review Board (IRB).
* Meet the Classification of Psoriatic Arthritis (CASPAR) criteria for PsA
* Participants must have a Body Mass Index (BMI) of 30kg/m^2
* Participants must be treated for PsA in accordance with guidelines
* Have not achieved MDA in PsA patients
* Have a minimum TJC > 1 and SJC > at baseline
* Eligible for GLP-1 agonist treatment in accordance with Food Drug Administration (FDA) labeling as determined by the investigator.

Exclusion Criteria:

* Any prior use of GLP-1 agonists
* Inability to provide informed consent
* Current participation in another PsA study
* Treatment initiation by GLP-1 agonists contraindicated by FDA
* Patients with hemoglobin A1c (HbA1c) > 10 at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2028-10-15 (Estimated)

PRIMARY OUTCOMES:
Change from the baseline Minimal Disease Activity (MDA) Scores at Week 12 and 24 with GLP-1 Agonists vs Nutrition Counseling | Week 12 and 24
  In order to meet Minimal Disease Activity (MDA) participants need to meet 5 of the 7 criteria: tender joint count less than or equal to 68 and greater than or equal to 1 (TJC68), swollen joint count less than or equal to 66 and greater than or equal to 1 (SJC66), psoriasis body surface area is less than or equal to 3%, patient pain Visual Analogue Scale (VAS) is less than or equal to 15mm, patient global disease activity VAS is less than or equal to 20mm, Health Assessment Questionnaire (HAQ) is less than or equal to 0.5 and tender entheseal points is less than or equal to 1. One of the outcomes of this study is to see how these scores change with the participants receiving a GLP-1 or nutrition counseling.
Proportion of Patients who Achieve Disease Activity in Psoriatic Arthritis (DAPSA) Remission with GLP-1 Agonists Vs. Nutrition Counseling at Week 12 and 24 | Week 12 and 24
  DASPA is a composite measure based on the summation of four variables: tender and swollen joints (TJC68, SJC66), C-reactive protein (CRP), Patient Global Assessment (PtGA) and Patient Pain both reported on a 0-100 mm VAS. DASPA classifications validated for PsA include Less than or equal to 4 (remission), greater than 4 but less than or equal to 14 is low disease activity. Greater than 14 but less than or equal to 28 is moderate disease activity and greater than 28 is high disease activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin/Froedtert Hosptial, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing at National/international conferences